CLINICAL TRIAL: NCT05688020
Title: Comparison Between Epinephrine Versus Tranexamic Acid Usage During Upper Gastrointestinal Tract Endoscopic Resection Procedures for the Reduction of Intraprocedural and Postprocedural Bleeding
Brief Title: Tranexamic Acid During Upper GI Endoscopic Resection Procedures
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 0118-22-ASF
Record Dates: First submitted 2023-01-05; First posted 2023-01-18 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Gastric Polyp; Gastric Neoplasm; Duodenal Neoplasms; Esophageal Neoplasms
MeSH Terms: conditions — Polyposis, Gastric; Stomach Neoplasms; Duodenal Neoplasms; Esophageal Neoplasms | interventions — Tranexamic Acid; Epinephrine

STUDY DESIGN:
Intervention Model Description: This study is designed as a prospective, double-blinded, controlled, non-inferiority pilot study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tranexamic acid (Experimental): During the ER procedure, de-identified injectate solution will be introduced. Study group: 9 ml of standart solution for injection [Consisit of: 6 ml indigo carmine + 500 ml succinylated gelatin 4% (Gelofusine; B. Braun, Crissier, Switzerland)] + 1 ml (100mg) of TXA (tranexamic acid).
  Interventions: Drug: Tranexamic acid
- Epinephrine (Active Comparator): During the ER procedure, de-identified injectate solution will be introduced. 9 ml of standart solution for injection [Consisit of: 6 ml indigo carmine + 500 ml succinylated gelatin 4% (Gelofusine; B. Braun, Crissier, Switzerland)] + 1 ml epinephrine 1:100,000 + 1 ml saline 0.9%.
  Interventions: Drug: Epinephrine injection

INTERVENTIONS:
Drug: Tranexamic acid — Tranexamic acid will be injected as part of the injectate during endoscopic resection.
  Other Names: Hexakapron
  Arms: Tranexamic acid
Drug: Epinephrine injection — Epinephrine will be injected as part of the standard injectate used during endoscopic resection.
  Other Names: Adrenaline
  Arms: Epinephrine

SUMMARY:
Endoscopic resection of gastrointestinal lesions may prevent cancer. However, resection is associated with adverse events such as bleeding. Tranexamic acid (TXA) is a synthetic derivative of lysine that exerts antifibrinolytic effects and may prevent bleeding. The investigators aim to evaluate the effect of local TXA on preventing intraprocedural and postprocedural bleeding in patients undergoing endoscopic mucosal resection (EMR) of upper gastrointestinal lesions.

DETAILED DESCRIPTION:
Endoscopic resection (ER) is an endoscopic technique used for the removal of sessile or flat neoplasms confined to the superficial layers (mucosa and submucosa) of the gastrointestinal (GI) tract.

This technique is not without risk, and clinically significant intraprocedural bleeding and post-ER bleeding remain the most frequently encountered serious adverse event.

The bleeding rate associated with ER varies for the different regions of the GI tract. This is most probably due to differences in the vascularity within the wall of the GI tract in each region.

Intraprocedural bleeding in the stomach and duodenum is more frequent and may be as high as 11.5% and 19.3%, respectively. Delayed bleeding has been reported at about 5% for these sites.

Management of bleeding is often resource intensive and may necessitate hospitalization, blood transfusion, and repeat intervention. Some techniques, such as soft coagulation with the tip of a snare; epinephrine injection; hemoclip placement or proton-pump inhibitor treatment, are used to decrease the risk of bleeding or treat active bleeding.

Diluted epinephrine, which causes vasoconstriction, is often added to the submucosal injection fluid because of the theoretical benefit of decreasing bleeding. However, epinephrine has a short time-of-action and for long procedures it requires multiple doses to be injected. This can result in systemic effects such as severe hypertension, ventricular tachycardia, and intestinal ischemia, and may also increase postprocedural pain and prolong patient observation after the procedure.

Tranexamic acid (TXA) is a synthetic derivative of lysine that exerts antifibrinolytic effects by inhibition of lysine binding sites on plasminogen molecules and therefore stabilizes the fibrin meshwork produced by secondary hemostasis. TXA was patented by Dr. S. Okamoto in 1957, and it was found to be significantly more potent than a precursor molecule known as epsilon-amino-caproic acid.

During the past few years, TXA has been 'rediscovered' and is currently used in many conditions that are associated with either overt or occult hemorrhage. It is one of the most frequently cited drugs in recent surgical publications involving nearly all surgical specialties.

After the CRASH-2 study which showed that administration of TXA to bleeding trauma patients within 3 hours of injury significantly reduced the risk of death due to bleeding and all-cause mortality without increasing the risk of vascular occlusive events, it has become an important part of trauma management.

It is also widely used in gynecological practice. Early treatment with TXA reduces death due to bleeding in women with post-partum hemorrhage, as well as total blood loss and transfusion requirements in hemorrhage after caesarean delivery. Therefore, TXA has been recommended by the WHO as part of postpartum hemorrhage management.

TXA is also commonly used in orthopedic surgery, either systemically or topically, to reduce excessive bleeding and transfusion requirements.

Other hemorrhagic conditions in which TXA has been shown effective are epistaxis, hemoptysis , endoscopic ear surgery , mastectomy, and hereditary hemorrhagic telangiectasia with bleeding.

Topical use of TXA may be more beneficial than systemic use as it may provide a higher drug concentration on the wound surface with negligible systemic concentrations. Most publications concerning topically administered TXA come from orthopedic literature where instilling TXA as a bolus into the joint reduces bleeding. Recently, a study revealed that intradermal injections of TXA in dermatological surgery reduces bleeding, especially in those on anticoagulant medications.

While TXA is an inhibitor of fibrinolysis, and therefore might theoretically increase the risk of thrombotic vascular events, most studies show no increased risk of thromboembolism. This finding has been consistent with all routes of TXA administration including IV, topical/intra-articular, and other routes.

The most frequently described contraindications to TXA administration include patients with histories of allergic reactions to TXA, seizures, and patients with acute renal failure or chronic kidney disease.

The investigators propose that the use of TXA in the injection gel during ER procedures will be as effective as epinephrine usage in reducing intraprocedural and postprocedural bleeding, while also decreasing the incidence of side effects including abdominal pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for endoscopic resection of a non-neoplastic and neoplastic lesions in the upper GI presenting to our tertiary academic center.
* Age > 18 years

Exclusion Criteria:

* patients with histories of allergic reactions to TXA
* history of seizures
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Intraprocedural bleeding | During procedure
  To compare the severity of intraprocedural bleeding between those receiving TXA and those receiving epinephrine.
Postprocedural bleeding | 2 weeks post-procedure
  To compare the severity of postprocedural bleeding between those receiving TXA and those receiving epinephrine.

SECONDARY OUTCOMES:
Side effects | 2 weeks post-procedure
  To compare the number and severity of occurrences of abdominal pain, tachycardia, and hypertension between those receiving TXA and those r receiving epinephrine.

CONTACTS AND LOCATIONS:
Overall Officials: Anton Bermont, MD, Principal Investigator — Assaf-Harofeh Medical Center
Locations (1):
- Shamir Medical Center, Be’er Ya‘aqov, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] ASGE Technology Committee; Hwang JH, Konda V, Abu Dayyeh BK, Chauhan SS, Enestvedt BK, Fujii-Lau LL, Komanduri S, Maple JT, Murad FM, Pannala R, Thosani NC, Banerjee S. Endoscopic mucosal resection. Gastrointest Endosc. 2015 Aug;82(2):215-26. doi: 10.1016/j.gie.2015.05.001. Epub 2015 Jun 12. PMID 26077453
- [Background] Park CH, Lee SK. Preventing and controlling bleeding in gastric endoscopic submucosal dissection. Clin Endosc. 2013 Sep;46(5):456-62. doi: 10.5946/ce.2013.46.5.456. Epub 2013 Sep 30. PMID 24143302
- [Background] Libanio D, Pimentel-Nunes P, Dinis-Ribeiro M. Complications of endoscopic resection techniques for upper GI tract lesions. Best Pract Res Clin Gastroenterol. 2016 Oct;30(5):735-748. doi: 10.1016/j.bpg.2016.09.010. Epub 2016 Sep 14. PMID 27931633
- [Background] Yang Z, Wu Q, Liu Z, Wu K, Fan D. Proton pump inhibitors versus histamine-2-receptor antagonists for the management of iatrogenic gastric ulcer after endoscopic mucosal resection or endoscopic submucosal dissection: a meta-analysis of randomized trials. Digestion. 2011;84(4):315-20. doi: 10.1159/000331138. Epub 2011 Nov 9. PMID 22075541
- [Background] Castro R, Libanio D, Pita I, Dinis-Ribeiro M. Solutions for submucosal injection: What to choose and how to do it. World J Gastroenterol. 2019 Feb 21;25(7):777-788. doi: 10.3748/wjg.v25.i7.777. PMID 30809079
- [Background] Watts G. Utako Okamoto. Lancet. 2016 Jun 4;387(10035):2286. doi: 10.1016/s0140-6736(16)30697-3. No abstract available. PMID 27308678
- [Background] Montroy J, Hutton B, Moodley P, Fergusson NA, Cheng W, Tinmouth A, Lavallee LT, Fergusson DA, Breau RH. The efficacy and safety of topical tranexamic acid: A systematic review and meta-analysis. Transfus Med Rev. 2018 Feb 19:S0887-7963(17)30151-7. doi: 10.1016/j.tmrv.2018.02.003. Online ahead of print. PMID 29567052